CLINICAL TRIAL: NCT00961870
Title: Effect of Radius Subjecting to Mechanical Loading on Alpha Motor Neuron Excitability
Brief Title: Effect of Radius on Alpha Motor Neuron Excitability
Acronym: ERAMNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ILHAN KARACAN, ILHAN KARACAN, Vakif Gureba Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VGEAH FTR-2
Record Dates: First submitted 2009-08-14; First posted 2009-08-19 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Osteoporosis
Keywords: bone; motor neuron excitability; forearm vibration; Mechanical Loading
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy postmenopausal women (Experimental): Forearm vibration will be applied in women without postmenopausal osteoporosis
  Interventions: Procedure: Forearm vibration
- Osteoporotic postmenopausal women (Experimental): Forearm vibration will be applied in women with postmenopausal osteoporosis
  Interventions: Procedure: Forearm vibration
- Healthy young adult women (Experimental): Forearm vibration will be applied in healthy young adult women
  Interventions: Procedure: Forearm vibration
- Healthy young adult men (Experimental): Forearm vibration will be applied in healthy young adult men
  Interventions: Procedure: Forearm vibration

INTERVENTIONS:
Procedure: Forearm vibration — Mechanical loading with forearm vibration will be applied right radius in all groups.
  Other Names: Cyclic mechanical loading

SUMMARY:
This study hypothesize that radius subjecting to mechanical loading may affect excitability of alpha motor neuron innervating muscle, based on its bone mineral density. If this hypothesis is valid, it can be firstly suggested that the relationship between bone mineral density and muscle strength is bidirectional.

A total of 80 voluntaries are planned to include in this study.

After forearm vibration is applied, bone mineral density (BMD) and bone mineral content (BMC) will be measured in all cases. Alpha motor neuron excitability (H/M ratio, recruitment), background muscle activity will be evaluated by electromyography at pre-treatment, post-treatment and, during treatment in cases.

Forearm vibration will be applied by forearm vibration device (FAV). FAV with mechanical loading will apply forearm. Cases will sit on armchair. Two intervals of FAV will be applied at a frequency of 45 Hz. Each interval will consist of 60 second of FAV followed by rest.

The right radius BMD and BMC will be evaluated by bone densitometer (GE-LUNAR DPX PRO).

Motor unite potentials at rest, Hoffman reflex, F response, M response will be measured by electromyography at right flexor carpi radialis. Medtronic Keypoint Portable 2 channel electromyography and Neurotrac ETS device will be used.

DETAILED DESCRIPTION:
It is usually reported that there is a parallelism between changes in the bone structure and function and the muscle structure and function. Sarcopenia is frequently observed in osteoporotic patients. Bone formation increases or bone resorption decreases with exercise.

To date, the effect of bone on the muscle activity is not investigated. One of the most important functions of bone bear mechanical loads include body weight. Bone must be strong enough to resist the mechanical loading. Mechanisms need to protect bone when bone is subject to excessive mechanical loading. These mechanisms may mainly focus on strengthening the bone and/or changing vectorial properties of mechanical loading applied bone.

The vectorial properties of mechanical loading applied bone may be controlled by muscle contractions. Bone contains wide mechanoreceptor net constructed by osteocytes. So,distribution of the mechanical loading on bone cross-sectional area is possible to perceive. It may be also possible that inappropriate distribution of mechanical loading on bone crosssectional area is optimized by muscle contractions. To get this regulation, there should be a mechanism that muscle activity is controlled by central nervous system based on mechanical loading distribution on bone cross-sectional area. We previously showed that bone can regulate muscle activity, based on its bone mineral density. According to this study result, it can be suggested there may exist a mechanism that bone sensing mechanical stimuli can send the signals to central nervous system and neuronally regulate muscle activity (bone myo-regulation reflex). (It is also well known that load-induced adaptive bone formation is neuronally regulated. Taken together, a general mechanism, bone reflex, may be defined that bone subjected to loading can neuronally regulate bone formation and muscle activity)

This study hypothesize that radius subjecting to mechanical loading may affect excitability of alpha motor neuron innervating muscle, based on its bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* females with postmenopausal osteoporosis (forearm BMD: T score <-2.0)
* females without postmenopausal osteoporosis (forearm BMD: T score >-1.0)
* healthy young adult females (forearm BMD normal)
* healthy young adult males (forearm BMD normal)
* cases with right handed patients in all groups

Exclusion Criteria:

* secondary osteoporosis
* neuropathy (central or peripheral)
* myopathy
* systemic diseases (arthritis, endocrine-metabolic diseases, bone diseases)
* professional sportswoman/sportsman
* subjects doing regular sports activities
* tendinopathy
* amputee, endoprosthesis, metal implants

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changing alpha motor neuron excitability | 1-2 months

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Vakif Gureba Training & Research Hospital
Locations (1):
- Vakif Gureba Training & Research Hospital, Istanbul, Turkey (Türkiye)